CLINICAL TRIAL: NCT02024503
Title: A Longitudinal Study of Multimodal Resonance Imaging in Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor of Radiology & Chair,Department of Radiology, Zhongda Hospital
Other Study IDs: 2013CB733803
Record Dates: First submitted 2013-12-25; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Stroke
Keywords: stroke; fMRI; DTI
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extraction of DNA from the blood of patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental group: Hospitalized patients with acute stroke.
- Control group: Healthy Volunteers.

SUMMARY:
Imaging of the ischaemic penumbra with a particular diffusion-weighted imaging (DWI)/ perfusion-weighted imaging (PWI) mismatch is a promising approach to the selection of patients with acute ischaemic stroke for trials of intervention. The investigators want to apply multimodal resonance imaging methods such as functional magnetic resonance imaging ( fMRI), diffusion tensor imaging (DTI), arterial spin labeling (ASL) to guide treatment and predict the prognosis of stroke.

ELIGIBILITY:
Inclusion Criteria:

Time from the onset of stroke till hospital within 24 hours. With clinical characteristics such as hemiplegia, headache. Willing and able to comply with the study procedures and provide written informed consent to participate in the study.

Patients must understand the nature of the study and give informed consent.

Exclusion Criteria:

The onset of stroke out of 24 hours. Pregnant women. Patients with intracranial metallic bodies from prior neurosurgical procedure, implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit or ventriculoperitoneal shunt.

Past history of seizures within one year or unexplained loss of consciousness. Family history of epilepsy.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with stroke and the some healthy volunteers recruited from community
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Functional recovery | Participants will be followed till die or lost to follow-up,an expected average of three year.

SECONDARY OUTCOMES:
Over survival | Participants will be followed till die or lost to follow-up,an expected average of three year
  Time from stenting to the day when the patients died or lost to the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gao-jun Teng, Ph.D,MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital,Southeast University, Nanjing, Jiangsu, China